CLINICAL TRIAL: NCT01859884
Title: Optimizing Kidney Transplant Patients' Informed Consent for Increased Risk Donors
Brief Title: Optimizing Kidney Transplant Informed Consent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Elisa Gordon, Principal Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STU00055356
Record Dates: First submitted 2013-05-20; First posted 2013-05-22 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: End-stage Kidney Disease
Keywords: Kidney transplantation; Increased risk donor kidneys; Kidney donation; Organ donation; Human Immunodeficiency Virus; Hepatitis B; Hepatitis C; Infectious disease; Disease transmission; Centers for Disease Control (CDC); Web-based intervention
MeSH Terms: conditions — Kidney Failure, Chronic; Acquired Immunodeficiency Syndrome; Hepatitis B; Hepatitis C; Communicable Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inform Me: web-based education tool (Experimental): Intervention will receive the standard of care, the Inform Me intervention, a post-test evaluation, and 1 week recall test.
  Interventions: Behavioral: Inform Me: web-based education tool
- Control Standard of Care (No Intervention): This group receives standard of care with a post test.

INTERVENTIONS:
Behavioral: Inform Me: web-based education tool — The purpose of Inform Me is to help kidney transplant candidates understand what kidneys from increased risk donors are and describes the risks and benefits of accepting and refusing a kidney from an increased risk donor. Increased risk donors are donors who engaged in behaviors that increase their chances of having: Human Immunodeficiency Virus, Hepatitis B Virus , Hepatitis C Virus. Inform Me focuses only on increased risk donor kidneys. Inform Me aims to prepare patients to make a decision with their transplant team to accept or to refuse a kidney from an increased risk donor. Inform Me does not try to convince patients to accept or refuse a kidney from increased risk donors.
  Arms: Inform Me: web-based education tool

SUMMARY:
The objective of this study is to evaluate kidney transplant candidates' comprehension about increased risk donor kidneys necessary for informed consent. We have developed a web-based tool that educates and assesses candidates' comprehension (Inform Me), as a supplement to current informed consent processes. We will then compare the effectiveness of the current informed consent processes supplemented by Inform Me, with the current consent processes alone for kidney transplant.

DETAILED DESCRIPTION:
The shortage of kidneys for kidney transplantation results in almost 10,000 deaths per year in the United States. One strategy to increase the number of available kidneys is to offer kidney transplant candidates kidneys that come from donors who have an increased risk of transmission of human immunodeficiency virus (HIV), Hepatitis B and Hepatitis C. Increased risk kidney donors are defined as those who have engaged in behaviors associated with an increased risk of HIV, Hepatitis B, and Hepatitis C, and comprise approximately 9% of all US deceased organ donors. The Organ Procurement and Transplantation Network policy mandated informed consent from recipients who accept increased risk kidneys. The objective of this study is to increase study participants' comprehension about increased risk donor kidneys necessary for informed consent. To accomplish this objective, we will develop a web-based tool that educates and assesses participants' comprehension (Inform Me), as a supplement to current informed consent processes. We will then compare the effectiveness of the current informed consent processes supplemented by Inform Me, with the current consent processes alone. The tool will utilize health information technology to deliver information about the definition of, risks, benefits, and alternatives to using increased risk donor kidneys via a web-based application. Computer adaptive learning will personalize information presented to each candidate according to his/her comprehension levels in interactive chapters to increase comprehension. Inform Me will facilitate nurses' primary role as patient educators.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* 21 years or older
* Kidney Transplant candidates eligible: 1) completed the first phase of transplant evaluation education, and 2) wait-listed patients expected to receive a transplant within the next 6 months, returning for re-evaluation.

Exclusion Criteria:

* No special classes of study participants, including fetuses, neonates, prisoners, institutionalized individuals, or other vulnerable populations will be included in the proposed study. Although pregnant women will be eligible for participation in the study, they are unlikely to be selected for kidney transplantation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Actual)
Dates: Start 2013-10; Primary Completion 2014-12 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Knowledge of increased risk donor kidney transplants | 1 week
  Assess knowledge of increased risk donor kidneys

SECONDARY OUTCOMES:
Willingness to accept an increased risk donor kidney transplant | 1 week
  Willingness to accept an increased risk donor kidney.

OTHER OUTCOMES:
Decisional conflict | 1 week
  Will measure difficulty in treatment decision-making.
Satisfaction with the informed consent process | 1 week
  Assess decision-making quality, decision satisfaction, and perception of information.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Gordon, PhD, MPH, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Northwestern Memorial Hospital, Chicago, Illinois

REFERENCES:
- [Derived] Gordon EJ, Sohn MW, Chang CH, McNatt G, Vera K, Beauvais N, Warren E, Mannon RB, Ison MG. Effect of a Mobile Web App on Kidney Transplant Candidates' Knowledge About Increased Risk Donor Kidneys: A Randomized Controlled Trial. Transplantation. 2017 Jun;101(6):1167-1176. doi: 10.1097/TP.0000000000001273. PMID 27463536